CLINICAL TRIAL: NCT01497548
Title: A Parallel-group, Double-blind, Placebo-controlled Study of Methylphenidate as an Add on Therapy for Mirtazapine in the Treatment of Major Depressive Disorder in Cancer Patients Under Palliative Care
Brief Title: Study of Methylphenidate as Add on Therapy in Depressed Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Ng Chong Guan, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCG001
Record Dates: First submitted 2011-02-24; First posted 2011-12-22 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: Depression
Keywords: Depression; cancer; methylphenidate; pharmacotherapy
MeSH Terms: conditions — Depression; Neoplasms | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate add on to Mirtazapine (Experimental): Methylphenidate add on to the usual treatment (Mirtazapine)
  Interventions: Drug: Methylphenidate
- Placebo add on to Mirtazapine (Placebo Comparator): Non active compund add on to the usual treatment (Mirtazapine)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate started at 5mg on morning (0800) and noon (1200) on day 1. Dose increased to 10mg on morning (0800) and noon (1200) on day 3; 15mg on morning and noon on day 6 depending on the clinical response. Similarly, the dose can be reduced to 5mg/day if patients are not able to tolerate a higher dose. The treatment continues until day 28.
  Other Names: Ritalin
  Arms: Methylphenidate add on to Mirtazapine
Drug: Placebo — Placebo given on morning (0800) and noon (1200)daily
  Other Names: Non active compound
  Arms: Placebo add on to Mirtazapine

SUMMARY:
Primary Objective To determine the efficacy of Methylphenidate as add on therapy to mirtazapine in the treatment of depression in cancer patients under palliative care Hypothesis Methyphenidate add on to mirtazapine treated subjects will show significant early reduction in (Montgomery Asberg Depression Rating Scale) MADRS between baseline and Day 3.

Secondary Objective

1. To determine the efficacy of Methylphenidate as add on therapy to mirtazapine in the treatment of anxiety in cancer patients under palliative care.

   Hypothesis Methyphenidate add on to mirtazapine treated subjects will show significant early reduction in anxiety score of HADS than Mirtazepine alone treated subjects between baseline and Day 3.
2. To determine the efficacy of Methylphenidate as add on therapy to mirtazapine in reducing distress in cancer patients under palliative care.

   Hypothesis Methyphenidate add on to mirtazapine treated subjects will show significant early reduction in distress score of distress thermometer than Mirtazepine alone treated subjects between baseline and Day 3.
3. To determine the efficacy of Methylphenidate as add on therapy to mirtazapine in improving function in cancer patients under palliative care.

   Hypothesis Methyphenidate add on to mirtazapine treated subjects will show increase in the (Eastern Cooperation Group performance status) ECOG score than Mirtazepine alone treated subjects between baseline and Day 3
4. To determine the efficacy of Methylphenidate as add on therapy to mirtazapine in reducing somatic complaints in cancer patients under palliative care.

Hypothesis Methyphenidate add on to mirtazapine treated subjects will show significant early reduction in the score of Numeric Rating Scale (NRS) for Pain and Visual Analogue Scale (VAS) for Fatigue than Mirtazapine alone treated subjects between baseline and Day 3.

DETAILED DESCRIPTION:
Background

Cancer remains one of the most feared illnesses and the diagnosis of cancer has huge psychological impact on the patients and their care-takers (Knobf, 2007). Depression is one the most common psychiatric sequella (Derogatis et al., 1983)2 and affects the quality of life, compliance to treatment, disease advancement, tolerability to pain and fatigue in cancer patients (Bennett et al., 2004; Sommerset, 2004; Green et al., 2009). However, it is likely that depression is under-recognized and under-treated in cancer patients (Kadan-Lottick et al., 2005).

Depressed feelings manifest in a spectrum ranging from normal sadness to a variety of mood disturbances and clinical presentations. It is challenging to differentiate clinical depression from "normal" emotional distress in cancer patients and the somatic symptoms such as fatigue, loss of appetite or weight, sleep difficulties, poor memory and concentration may mirror the physiological symptoms caused by cancer or its treatment (McDaniel and Musselman, 1995; Masie and Popkin, 1998; Cochinov, 2001; Jesse et al., 2008). This complicates the diagnosis of depression in cancer patients (McDaniel and Musselman, 1995; Masie and Popkin, 1998; Cochinov, 2001; Pasquini and Biond, 2007; Jesse et al., 2008).

Many studies have investigated the prevalence of depression in cancer in the past decades. A previous review by Mc Daniel et al, reported a prevalence of major depression ranging from 4.8% to 9.2% based on studies using standardized diagnostic interviews on cancer outpatients. Prevalence rates were higher in the admitted cancer patients (8% for Major Depression and 15% to 36% for all depressive disorders)(McDaniel and Musselman, 1995). A preliminary systematic review on the prevalence of depression in cancer patients was conducted by the investigator of this study. It showed that major depressive disorder was as high as 10.8% in cancer patients based on structured clinical interview.

In addition to the high prevalence, uncertainty exists with respect to the optimal treatment of depression in cancer. Although a huge number of studies investigated the efficacy of pharmacotherapy for depression in general population, the number of randomized, controlled trials of antidepressants on depression in cancer patient conducted is limited(Challman and Lipsky, 2000; Raison and Miller, 2003). A comprehensive systematic review looking into the effectiveness and tolerability of antidepressant treatment in depressed cancer patients was performed and published by Rodin et al in 2007. Although 7 trials were identified, the authors commented that the number of positive randomized trials was limited and there is a need for more rigorous studies on other newer agents or alternative treatment option (Raison and Miller, 2003). The preliminary systematic review conducted by the investigator of this study also came to the same conclusion.

Psychostimulants such as methylphenidate have been proposed for the treatment of depressed patients because of their rapid onset of action (Masand and Tesar, 1995; Challman and Lipsky, 2000; Rozans et al., 2002; Kaminski and Sjogren, 2007). They may have antidepressant effects and may be advantageous due to the rapid onset of action (Candy et al., 2008). Some studies suggest they provide a safe and effective treatment of depression in cancer patients (Masand and Tesar, 1995) and alleviates opioid induced somnolence, improve cognitive function and ameliorate pain in cancer patients. Another potential advantage of the use of psychostimulant in the cancer patients is the ability to improve multiple somatic symptoms irrespective of the etiology (Vigano et al., 1995). However, the number of studies looking into the efficacy of psychostimulant in improving depressive mood in cancer is limited.

Five studies were identified from the review conducted by the investigator of this study. Although they showed positive result on the use of methylphenidate in depressed cancer patients, they were open-label and without control group. There is only one double blind, randomised placebo controlled study on the use of methylphenidate in cancer patients which was published in French language (Laval, 2008).Considering the lack of randomized controlled trial on the topic, the need of study on the efficacy and tolerability of psychostimulant such as methylphenidate as an add on therapy of depression in cancer patients is inevitably needed.

Primary Objective To determine the efficacy of Methylphenidate as add on therapy to mirtazapine in the treatment of depression in cancer patients

Secondary Objective

1. To determine the efficacy of Methylphenidate as add on therapy to mirtazapine in the treatment of anxiety in cancer patients.
2. To determine the efficacy of Methylphenidate as add on therapy to mirtazapine in reducing distress in cancer patients.
3. To determine the efficacy of Methylphenidate as add on therapy to mirtazapine in improving function in cancer patients.
4. To determine the efficacy of Methylphenidate as add on therapy to mirtazapine in reducing somatic complaints in cancer patients.

Study Design

Design An open label, parallel group, placebo controlled study on methylphenidate as add on therapy to mirtazapine.

Procedure Subjects will be male or female with current diagnosis of cancer of any types and DSM-IV diagnoses of major depressive disorder. They are identified from the oncology, surgical and palliative clinics and wards. Depressive symptoms will be measured at screening with the MADRS.

Sixty (120) subjects will be recruited and started on the mirtazapine 30mg at night. They will be then randomized to one of two groups (60 subjects per group): Methylphenidate or Placebo as add on therapy. All treatment will be initiated after screening and continued for 28 days of outpatient or inpatient treatment. Efficacy evaluation will be take place at baseline, day 3, day 6, 9, 14, 21 and day 28.

At the end of the 28 days, the continuation of treatment will be depends on the investigator's clinical judgment and End of Medication Evaluation will be perform. Every effort will be made to continue to evaluate all subjects who are randomized even if they decide to discontinue the medication.

Project Timetable The project will take 2 years. The plan is to randomize 2 subjects per week, taking about 15 month to acquire 120 subjects. All subjects will have completed study drug treatments before 18 months have elapsed. Follow-up evaluations will be completed 2 year from the start of the project.

Primary Study Endpoints

The primary endpoints to be measured in this study are:

- MADRS at the baseline, Day 3, 6, 9, 14, 21 and 28.

Secondary Study Endpoints

The secondary endpoints to be measured are:

* Anxiety with HADS at baseline, Day 3, 6, 9, 14, 21 and 28
* Distress score with distress thermometer at baseline, Day 3, 6, 9, 14, 21 and 28
* Karnofsky Scale at the baseline, Day 3, 6, 9, 14, 21 and 28
* Numeric Rating Scale (NRS) for Pain at the baseline, Day 3, 6, 9, 14, 21 and 28
* Visual Analogue Scale (VAS) for Fatigue at the baseline, Day 3, 6, 9, 14, 21 and 28

Primary Safety Endpoints The primary safety endpoint will be measurement and collection of any serious adverse event that occurs from initial study treatment through and including 14 days after cessation of study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged >18 years.
2. Current DSM IV diagnosis of Major Depressive Disorder.
3. Under palliative care.
4. Confirmed diagnosis of cancer.
5. Not on any antidepressants

Exclusion Criteria:

1. Clinical significant abnormal laboratory values.
2. Clinically significant abnormal ECG.
3. Documented history of other psychiatric diagnosis (schizophrenia, bipolar disorder, organic brain disorder, dementia etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-09 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
depressive symptoms | 3 to 28 days
  measured with Montgomery-Åsberg Depression Rating Scale

SECONDARY OUTCOMES:
Distress level | 3 to 28 days
  Measured with distress thermometer

CONTACTS AND LOCATIONS:
Overall Officials: Chong Guan Ng, MBBS, MPM, Principal Investigator — Department of Psychological Medicine, University Malaya Medical Centre
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Knobf MT. Psychosocial responses in breast cancer survivors. Semin Oncol Nurs. 2007 Feb;23(1):71-83. doi: 10.1016/j.soncn.2006.11.009. PMID 17303518
- [Background] Derogatis LR, Morrow GR, Fetting J, Penman D, Piasetsky S, Schmale AM, Henrichs M, Carnicke CL Jr. The prevalence of psychiatric disorders among cancer patients. JAMA. 1983 Feb 11;249(6):751-7. doi: 10.1001/jama.249.6.751. PMID 6823028
- [Background] Somerset W, Stout SC, Miller AH, Musselman D. Breast cancer and depression. Oncology (Williston Park). 2004 Jul;18(8):1021-34; discussion 1035-6, 1047-8. PMID 15328896
- [Background] Bennett B, Goldstein D, Lloyd A, Davenport T, Hickie I. Fatigue and psychological distress--exploring the relationship in women treated for breast cancer. Eur J Cancer. 2004 Jul;40(11):1689-95. doi: 10.1016/j.ejca.2004.03.021. PMID 15251158
- [Background] Green CR, Montague L, Hart-Johnson TA. Consistent and breakthrough pain in diverse advanced cancer patients: a longitudinal examination. J Pain Symptom Manage. 2009 May;37(5):831-47. doi: 10.1016/j.jpainsymman.2008.05.011. Epub 2008 Dec 2. PMID 19054648
- [Background] Kadan-Lottick NS, Vanderwerker LC, Block SD, Zhang B, Prigerson HG. Psychiatric disorders and mental health service use in patients with advanced cancer: a report from the coping with cancer study. Cancer. 2005 Dec 15;104(12):2872-81. doi: 10.1002/cncr.21532. PMID 16284994
- [Background] Massie, M.J., Popkin, M.K. Depressive Disorders. In: Holland, J.C. (Eds), Psycho-oncology. Oxford University Press, NY 1998; 518-519.
- [Background] Chochinov HM. Depression in cancer patients. Lancet Oncol. 2001 Aug;2(8):499-505. doi: 10.1016/S1470-2045(01)00456-9. PMID 11905726
- [Background] Fann JR, Thomas-Rich AM, Katon WJ, Cowley D, Pepping M, McGregor BA, Gralow J. Major depression after breast cancer: a review of epidemiology and treatment. Gen Hosp Psychiatry. 2008 Mar-Apr;30(2):112-26. doi: 10.1016/j.genhosppsych.2007.10.008. PMID 18291293
- [Background] McDaniel JS, Musselman DL, Porter MR, Reed DA, Nemeroff CB. Depression in patients with cancer. Diagnosis, biology, and treatment. Arch Gen Psychiatry. 1995 Feb;52(2):89-99. doi: 10.1001/archpsyc.1995.03950140007002. PMID 7848055
- [Background] Pasquini M, Biondi M. Depression in cancer patients: a critical review. Clin Pract Epidemiol Ment Health. 2007 Feb 8;3:2. doi: 10.1186/1745-0179-3-2. PMID 17288583
- [Background] Challman TD, Lipsky JJ. Methylphenidate: its pharmacology and uses. Mayo Clin Proc. 2000 Jul;75(7):711-21. doi: 10.4065/75.7.711. PMID 10907387
- [Background] Raison CL, Miller AH. Depression in cancer: new developments regarding diagnosis and treatment. Biol Psychiatry. 2003 Aug 1;54(3):283-94. doi: 10.1016/s0006-3223(03)00413-x. PMID 12893104
- [Background] Rodin G, Lloyd N, Katz M, Green E, Mackay JA, Wong RK; Supportive Care Guidelines Group of Cancer Care Ontario Program in Evidence-Based Care. The treatment of depression in cancer patients: a systematic review. Support Care Cancer. 2007 Feb;15(2):123-36. doi: 10.1007/s00520-006-0145-3. Epub 2006 Oct 21. PMID 17058100
- [Background] Rozans M, Dreisbach A, Lertora JJ, Kahn MJ. Palliative uses of methylphenidate in patients with cancer: a review. J Clin Oncol. 2002 Jan 1;20(1):335-9. doi: 10.1200/JCO.2002.20.1.335. PMID 11773187
- [Background] Marek Kaminski, Per Sjogren. The Use of psychostimulants in palliative and supportive treatment of cancer patients. Advances in Palliative Medicine 2007; 6: 23-31.
- [Background] Masand PS, Tesar GE. Use of stimulants in the medically ill. Psychiatr Clin North Am. 1996 Sep;19(3):515-47. doi: 10.1016/s0193-953x(05)70304-x. PMID 8856815
- [Background] Candy M, Jones L, Williams R, Tookman A, King M. Psychostimulants for depression. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD006722. doi: 10.1002/14651858.CD006722.pub2. PMID 18425966
- [Background] Vigano A, Watanabe S, Bruera E. Methylphenidate for the management of somatization in terminal cancer patients. J Pain Symptom Manage. 1995 Feb;10(2):167-70. doi: 10.1016/0885-3924(94)00080-5. PMID 7730689
- [Background] Laval G, Paris A. [Methylphenidate in palliative care in cancer patient: a double-blind randomised trial versus placebo]. Bull Cancer. 2008 Feb;95(2):241-6. doi: 10.1684/bdc.2008.0581. French. PMID 18304907
- [Derived] Ng CG, Boks MP, Roes KC, Zainal NZ, Sulaiman AH, Tan SB, de Wit NJ. Rapid response to methylphenidate as an add-on therapy to mirtazapine in the treatment of major depressive disorder in terminally ill cancer patients: a four-week, randomized, double-blinded, placebo-controlled study. Eur Neuropsychopharmacol. 2014 Apr;24(4):491-8. doi: 10.1016/j.euroneuro.2014.01.016. Epub 2014 Jan 20. PMID 24503279